CLINICAL TRIAL: NCT00247949
Title: The Accuracy of Non-invasive Continuous Carbon Dioxide Monitoring by the Sentec V-Sign Digital Monitor System
Brief Title: Accuracy of Non-invasive Continuous CO2-Monitoring
Status: Terminated | Type: Observational
Why Stopped: We had got enough data, therefore we stopped the study and published the data.
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: SenTec AG, Ringstrasse 39, CH-4106 Therwil (Unknown)
Responsible Party: Dr. D. Bolliger, MD
Other Study IDs: 52/04
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Blood Gas Monitoring, Transcutaneous
Keywords: carbon dioxide; monitoring; major surgery; repeated blood gas testing; carbon dioxide monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Arterial carbon dioxide partial pressure (PaCO2) is an essential indicator of ventilation and respiratory function. It is routinely tested invasively by arterial blood gas analysis (ABGA) but recently developed miniaturized carbon dioxide tension sensors promise non-invasive and continuous transcutaneous PCO2 (PtcCO2) monitoring. We, the researchers at University Hospital, Basel, Switzerland, determined the accuracy of two PtcCO2 monitors (TOSCA 500 with Sensor 92, Linde Medical Sensors AG, Basel; and Sentec Digital Monitor with V-Sign Sensor, Sentec AG, Therwil) for measurement of single values and trends in PaCO2 in critically ill patients, using ABGA as a reference.

DETAILED DESCRIPTION:
Measurement of SO2 is used in nearly every patient receiving anesthesia or sedation, whereas monitoring of pCO2 is important in patients during and shortly after major surgery and in critically ill patients. But measurement of pCO2 requires arterial blood sampling and laboratory testing. Non-invasive monitors for continuous assessment of arterial pCO2 have been developed but their accuracy and feasibility were insufficient to make them useful in the clinical setting. Recently, a new digital system for continuous and non-invasive monitoring of arterial pCO2 and SO2 has been introduced (SenTec Digital Monitor System, SenTec AG, Therwil, Switzerland). This present study has been designed to evaluate the accuracy of the SenTec V-SignTM monitoring system for measuring pCO2 in comparison with repeated arterial blood gas testing in the operation room and in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with clinical indication of repeated arterial blood gas analyses

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgery in general anesthesia and with clinical indication for repeated arterial blood gas sampling
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2004-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bolliger, Dr., Principal Investigator — Department of Anaesthesia University Hospital Basel
Locations (1):
- University Hospital, Basel, CH, Switzerland